CLINICAL TRIAL: NCT05112029
Title: Metabolic Profile and Adipokine Levels in Young Hyperandrogenemic Females
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Sponsor
Other Study IDs: ADIP-AN
Record Dates: First submitted 2021-10-14; First posted 2021-11-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Hyperandrogenism; Obesity; Metabolic Disease; Metabolic Syndrome
MeSH Terms: conditions — Hyperandrogenism; Obesity; Metabolic Diseases; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Deep frozen plasma and serum.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Assessement of basic metabolic profile and adipokine levels in young hyperandrogenemic females.

ELIGIBILITY:
Inclusion Criteria:

* hyperandrogenemia
* informed consent to participate
* female sex
* age 18-40 years old

Exclusion Criteria:

* male sex
* no consent given

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Hyperandrogenemic females admitted for additional assessment due to medical reasons.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-09-22 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Basic metabolic profile. | Day of blood testing - no further assessment planned (observational study).
  Serum lipids, uric acid, fasting glucose and insulin.
Adipokines. | Day of blood testing - no further assessment planned (observational study).

CONTACTS AND LOCATIONS:
Overall Officials: Renata Świątkowska-Stodulska, MD PhD, Study Director — Medical University of Gdansk; Agata Berlińska, MD, Principal Investigator — Medical University of Gdansk
Locations (1):
- Department of Endocrinology and Internal Medicine, Medical University of Gdansk, Gdansk, Poland